CLINICAL TRIAL: NCT03728205
Title: A Pilot Study On The Effect Of Yoga On Fatigue, And Stress Levels In Solid Tumor Cancer Patients Undergoing Active Radiation Therapy
Brief Title: Yoga for Solid Tumor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UPCC 13918; 831417 (Other: Penn Medicine)
Record Dates: First submitted 2018-10-29; First posted 2018-11-02 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational (Experimental): All 10 pilot subjects will be taking yoga
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — Twice weekly yoga sessions for 12 weeks

SUMMARY:
The purpose of this study is to ascertain the effect of yoga interventions on radiation-related fatigue, and stress in cancer patients with stage I and II solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Stage I and II Cancer patients with solid tumors undergoing RT for 4-8 weeks (external beam radiation).
2. Patients of age >18, and all races will be included in the study.
3. All patients must sign an informed consent form approved for this purpose by the Institutional Review Board (IRB) of the University of Pennsylvania.
4. Patients must be English speaking.
5. Patients must be able to attend the schedule classes.

   Exclusion Criteria:
6. Patients with medical restrictions that may interfere with or prevent them from taking part in the yoga interventions per their physician orders.
7. Patients with metastatic disease.
8. Active smokers. Smoking may interfere with relaxation and breathing modalities of the yoga interventions. (Self-reporting smokers that have been smoke free for 6 months may be included)
9. Patients who currently practice or have recently practiced yoga (had not taken a yoga class on a regular bases in the last 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
The feasibility of implementing Eischens yoga interventions for solid tumor cancer patients undergoing radiation therapy. This will be measured by the success rate of recruitment and retention for 10 subjects. | 12 months
  Feasibility

SECONDARY OUTCOMES:
Effects on fatigue | 12 months
  Examine the effect of yoga on cancer and radiation related fatigue during radiation therapy. We will use the BFI results both before, during and after radiation therapy.
Effects on Stress Level | 12 Months
  Examine the effect of yoga on cancer and radiation related fatigue during radiation therapy. We will use the NCCN Distress thermometer results both before, during and after radiation therapy.

OTHER OUTCOMES:
Long Term | 17 months
  Examine the long term effect of yoga to be tested at the 6 months post radiation visit. We will use the BFI and distress thermometer to see if any positive results during yoga are sustained to the 6 month follow up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided